CLINICAL TRIAL: NCT01484015
Title: Prolonged Infusion Compared to Standard Infusion Cefepime as Empiric Treatment of Febrile Neutropenia: A Pilot Study
Brief Title: Prolonged or Standard Infusion of Cefepime Hydrochloride in Treating Patients With Febrile Neutropenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015247; NCI-2011-02422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 02110 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-10-21; First posted 2011-12-02 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Adult Acute Lymphoblastic Leukemia; Adult Acute Myeloid Leukemia; Adult Burkitt Lymphoma; Adult Diffuse Large Cell Lymphoma; Adult Diffuse Mixed Cell Lymphoma; Adult Diffuse Small Cleaved Cell Lymphoma; Adult Hodgkin Lymphoma; Adult Immunoblastic Large Cell Lymphoma; Adult Lymphoblastic Lymphoma; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Breast Cancer; Chronic Eosinophilic Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Cutaneous T-cell Non-Hodgkin Lymphoma; Disseminated Neuroblastoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3 Follicular Lymphoma; Malignant Testicular Germ Cell Tumor; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Multiple Myeloma; Mycosis Fungoides/Sezary Syndrome; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neutropenia; Nodal Marginal Zone B-cell Lymphoma; Ovarian Epithelial Cancer; Ovarian Germ Cell Tumor; Plasma Cell Neoplasm; Poor Prognosis Metastatic Gestational Trophoblastic Tumor; Primary Myelofibrosis; Prolymphocytic Leukemia; Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Breast Neoplasms; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Multiple Myeloma; Mycosis Fungoides; Sezary Syndrome; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neutropenia; Carcinoma, Ovarian Epithelial; Neoplasms, Plasma Cell; Primary Myelofibrosis; Leukemia, Prolymphocytic | interventions — Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (standard infusion) (Experimental): Patients receive cefepime hydrochloride IV over 30 minutes.
  Interventions: Drug: cefepime hydrochloride
- Arm II (prolonged infusion) (Experimental): Patients receive cefepime hydrochloride IV over 3 hours. Treatment repeats every 8 hours.
  Interventions: Drug: cefepime hydrochloride

INTERVENTIONS:
Drug: cefepime hydrochloride — Given IV
  Other Names: cefepime; Maxipime

SUMMARY:
This randomized pilot clinical trial studies how well giving prolonged infusion compared to standard infusion of cefepime hydrochloride works in treating patients with febrile neutropenia. Giving cefepime hydrochloride over a longer period of time may be more effective than giving cefepime hydrochloride over the standard time.

DETAILED DESCRIPTION:
OBJECTIVES:

I. The objective of this study is to describe outcomes associated with prolonged infusion (3 hours) compared to standard infusion (30 minutes) cefepime (cefepime hydrochloride) among patients being treated empirically for febrile neutropenia.

OUTLINE: Patients are randomized 1 of 2 treatment arms.

All patients receive cefepime hydrochloride intravenously (IV) over 30 minutes as their first dose.

ARM I: Patients receive cefepime hydrochloride intravenously (IV) over 30 minutes.

ARM II: Patients receive cefepime hydrochloride IV over 3 hours. Treatment repeats every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count < 500 cells/mm^3 or < 1000 cells/mm^3 with a predicted decrease to < 500 cells/mm^3
* Temperature > 38.0 degrees Celsius
* Received chemotherapy or stem-cell transplant as treatment for malignancy or myelodysplastic syndrome (MDS)
* Cefepime prescribed at a dose of 2 grams IV every 8 hours

Exclusion Criteria:

* Allergy to a cephalosporin antibiotic
* Estimated creatinine clearance < 50 milliliters/minute
* Concurrent anti-gram negative antimicrobials
* Diagnostic criteria suggestive of sepsis
* Circumstances which may make 3 hour infusion impractical
* Solid tumor malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Defervescence (without hypothermia) | 72 hours
  Comparison between groups will be done using the chi square test. T-tests will be used for continues variables. Survival data will be estimated using the Kaplan-Meier method, with the formal test of group comparisons done using Cox's Proportional Hazards Model.

SECONDARY OUTCOMES:
Clinical success or failure | approximately 24 days
Need for additional antimicrobials | approximately 24 days
Mortality (in-house) | approximately 24 days
Time to defervescence | approximately 24 days
Hospital length of stay | approximately 24 days
Successful treatment of baseline infection | approximately 24 days

CONTACTS AND LOCATIONS:
Overall Officials: John Williamson, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States